CLINICAL TRIAL: NCT00103558
Title: A Phase I/II Study of Lumiliximab in Combination With Fludarabine, Cyclophosphamide, and Rituximab in Subjects With Relapsed Chronic Lymphocytic Leukemia
Brief Title: Lumiliximab in Combination With FCR in Subjects With Relapsed Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 152-30
Record Dates: First submitted 2005-02-10; First posted 2005-02-11 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — lumiliximab; Receptors, Fc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lumiliximab with FCR — Dose, schedule, and duration specified in protocol

SUMMARY:
This is an open label, Phase I/II, dose escalation research study of an investigational product called lumiliximab, given with FDA (Food and Drug Administration) approved products fludarabine, cyclophosphamide, and rituximab (FCR). The study duration is 17 visits over 42 months or until your disease progresses and you require additional CLL therapy. The total duration of participation in the study will be approximately 4 years, however your disease status will be followed indefinitely (forever).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Diagnosis of B-cell CLL by International Workshop on CLL (IWCLL) response criteria
* Relapsed CD23+ B-cell CLL
* Rai Stage III or IV, or Rai Stage I or II if determined to have disease progression as evidenced by rapid doubling or peripheral lymphocyte count, progressive lymphadenopathy, progressive splenomegaly, or B symptoms
* Prestudy WHO Performance Status less than or equal to 2
* Signed, written Institutional Review Board (IRB)-approved informed consent
* Men & women of reproductive potential must agree to follow accepted birth control methods during treatment for 3 months after completion of treatment
* Acceptable liver function: Bilirubin less than or equal to 2.0 mg/dL (26 µmol/L), AST (SGOT) &/or ALT (SGPT) less than or equal to 2 times upper limit of normal
* Acceptable hematologic status: Platelet count less than or equal to 50 x 10^9/L, ANC less than or equal to 1 x 109/L
* Acceptable renal function: Serum creatinine less than or equal to 1.5 times upper limit of normal

Exclusion Criteria:

* Subjects who did not respond to prior FCR therapy (relapsed within 6 months of the last dose).
* Cancer radiotherapy, radioimmunotherapy, biological therapy, chemotherapy, or other investigational therapy within 4 weeks prior to Study Day 1
* Previous exposure to lumiliximab or other anti-CD23 antibodies
* Subjects who have had a prior allogenic bone marrow transplant (BMT) or autologous BMT or peripheral stem-cell transplant (PBSCT)
* Known infection with HIV, hepatitis B, or hepatitis C
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* Transformation to aggressive B-cell malignancy (e.g., larger B-cell lymphoma, Richter's Syndrome, or prolymphocyte leukemia (PLL)
* Subjects with secondary malignancy requiring active treatment (except hormonal therapy)
* Subjects with medical conditions currently requiring long-term use (less than 1 month) of systemic corticosteroids
* Serious nonmalignant disease or laboratory abnormality, which, in the opinion of the investigator &/or sponsor, would compromise protocol objectives
* Active uncontrolled bacteria, viral, or fungal infections
* New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months prior to Study Day 1, unstable arrhythmia, or evidence of ischemia on ECG within 14 days prior to Study Day 1
* Seizure disorders requiring anticonvulsant therapy
* Severe chronic obstructive pulmonary disease with hypoxemia
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Study Day 1
* Clinically active autoimmune disease
* Subjects with a history of fludarabine-induced autoimmune cytopenia
* Pregnant or currently breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-03; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile | monthly until month 12, then every 3 months for 24 months, then every 6 months until month 48

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of lumiliximab and rituximab | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- United States (5):
  - Research Site, Birmingham, Alabama
  - Research Site, San Diego, California
  - Research Site, Baltimore, Maryland
  - Research Site, Columbus, Ohio
  - Research Site, Houston, Texas

REFERENCES:
- [Background] Pathan NI, Chu P, Hariharan K, Cheney C, Molina A, Byrd J. Mediation of apoptosis by and antitumor activity of lumiliximab in chronic lymphocytic leukemia cells and CD23+ lymphoma cell lines. Blood. 2008 Feb 1;111(3):1594-602. doi: 10.1182/blood-2007-03-082024. Epub 2007 Nov 21. PMID 18032710
- [Background] Byrd JC, O'Brien S, Flinn IW, Kipps TJ, Weiss M, Rai K, Lin TS, Woodworth J, Wynne D, Reid J, Molina A, Leigh B, Harris S. Phase 1 study of lumiliximab with detailed pharmacokinetic and pharmacodynamic measurements in patients with relapsed or refractory chronic lymphocytic leukemia. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4448-55. doi: 10.1158/1078-0432.CCR-06-1463. PMID 17671129
- [Derived] Byrd JC, Kipps TJ, Flinn IW, Castro J, Lin TS, Wierda W, Heerema N, Woodworth J, Hughes S, Tangri S, Harris S, Wynne D, Molina A, Leigh B, O'Brien S. Phase 1/2 study of lumiliximab combined with fludarabine, cyclophosphamide, and rituximab in patients with relapsed or refractory chronic lymphocytic leukemia. Blood. 2010 Jan 21;115(3):489-95. doi: 10.1182/blood-2009-08-237727. Epub 2009 Oct 20. PMID 19843887